CLINICAL TRIAL: NCT02543892
Title: Phase 1-2 Safety and Immunogenicity Study of PATH-wSP in Kenyan Adults and Toddlers
Brief Title: A Study of a Vaccine for Pneumonia in Adults and Toddlers in Kenya
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-040
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Pneumonia
Keywords: Vaccine
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Adult 0.6mg PATH-wSP (Experimental): Two 0.6 mg doses of PATH-wSP with a 28 day interval between doses
  Interventions: Biological: PATH-wSP
- Adult Placebo Low Dose (Placebo Comparator): Two injections of normal saline with a 28 day interval between injections
  Interventions: Biological: Placebo
- Adult 1.0 mg PATH-wSP (Experimental): Two 1 mg doses of PATH-wSP with a 28 day interval between doses
  Interventions: Biological: PATH-wSP
- Adult Placebo High Dose (Placebo Comparator): Two injections of normal saline with a 28 day interval between injections
  Interventions: Biological: Placebo
- Toddler 0.6mg PATH-wSP (Experimental): Two 0.6 mg doses of PATH-wSP with a 28 day interval between doses
  Interventions: Biological: PATH-wSP
- Toddler Placebo Low Dose (Placebo Comparator): Two injections of normal saline with a 28 day interval between injections
  Interventions: Biological: Placebo
- Toddler 1.0 mg PATH-wSP (Experimental): Two 1 mg doses of PATH-wSP with a 28 day interval between doses
  Interventions: Biological: PATH-wSP
- Toddler Placebo High Dose (Placebo Comparator): Two injections of normal saline with a 28 day interval between injections
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PATH-wSP — Streptococcus pneumoniae Whole Cell Vaccine, Inactivated and Adsorbed to Aluminum Hydroxide
  Arms: Adult 0.6mg PATH-wSP; Adult 1.0 mg PATH-wSP; Toddler 0.6mg PATH-wSP; Toddler 1.0 mg PATH-wSP
Biological: Placebo — Normal Saline
  Arms: Adult Placebo High Dose; Adult Placebo Low Dose; Toddler Placebo High Dose; Toddler Placebo Low Dose

SUMMARY:
This study aimed to determine whether PATH-wSP, a vaccine against a germ that causes pneumonia, is safe and induces immune responses in adults and toddlers. The study vaccine was compared to placebo. First adults received 2 injections of a lower dose of the vaccine or placebo, 28 days apart. Since the lower dose was considered safe, a higher dose was tested. Once the safety was established in adults the lower and higher dose was tested in toddlers, starting with the lower dose and then the higher dose.

DETAILED DESCRIPTION:
S. pneumoniae whole cell vaccine (SPWCV) is a vaccine candidate made from whole unencapsulated pneumococcal cells and adsorbed to aluminum hydroxide adjuvant (Alum). After adsorption of the Alum to SPWCV, the vaccine is referred to as PATH-wSP. PATH-wSP has been previously tested in Phase 1/2 studies in healthy US adults (VAC-002), and in healthy Kenyan adults and toddlers (VAC-010) and showed a favorable safety, tolerability, and immunogenicity profile. The SPWCV and Alum used in previous Phase 1/2 trials were supplied separately in a two-vial configuration; the SPWCV was manufactured at Walter Reed Army Institute of Research and the Alum at Instituto Butantan. A single-vial formulation of PATH wSP, an adsorbed suspension of SPWCV and Alum, has now been manufactured by PT Bio Farma, Indonesia. The purpose of this study was to assess the safety and tolerability of this new formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are 18 to 40 years old, or toddlers who are 12 to 19 months old.
* Must provide voluntary written/thumb-printed informed consent
* Must comply with study requirements and procedures.
* Must have an identifiable place of residence to allow home visits, and a consistent means of telephone contact
* Must be resident in the study area with no plans to travel outside the study area during the study
* Must be willing to not take herbal or other local traditional medications within 28 days of randomization and during the course of the study
* Adult female subjects must have a negative serum pregnancy test at screening and urine pregnancy test prior to each vaccination
* Toddlers must have been born full-term, and have a mid-upper arm circumference > 11.5 cm at the time of enrollment.
* Toddlers must have completed their Kenyan infant EPI schedule through 9 months including 1 birth dose of BCG, 3 doses of DTwPHibHep, 3 doses of OPV (birth dose is not required), 3 doses of PCV, and 1 dose of measles vaccine

Exclusion Criteria:

* Use of any investigational or nonregistered drug within 90 days of enrollment
* Use of any potentially hepatotoxic drug
* Receipt of any licensed vaccine within 14 days of administration of study vaccine.
* Chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or hematological functional abnormality or major congenital defects or illness that requires medical therapy, based on medical history or clinical assessment
* History of anaphylactic shock
* History of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines
* History of immunosuppression or immunodeficiency, inclusive of human immunodeficiency virus (HIV) infection by medical history (including that of an enrolled toddler's mother) or by HIV testing at screening
* Evidence of active hepatitis infection (B or C) by serologic testing at screening.
* Any screening laboratory test (chemistry or hematology) or vital sign measurement with toxicity grade ≥ 1
* Acute illness (moderate or severe) and/or fever (axillary temperature ≥ 37.5°C)
* Positive test for malaria (blood film) at screening that remains positive post treatment when retested prior to vaccination
* Disorders that require chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within the past 6 months prior to the administration of the study vaccine.
* Administration of immunoglobulins and/or any blood products within the 6 months preceding enrollment in the study
* Known disturbance of coagulation or other blood disorder (e.g., thalassemia, sickle cell disease, thrombocytopenia, disorders of the lymphocytes, severe anemia at birth) in adult subject or in self/first-degree relative of toddler subject; or receipt of anticoagulants in the past three weeks (aspirin as needed and nonsteroidal anti-inflammatory drugs are acceptable)
* History of meningitis, seizures or any neurological disorder (all participants) or major psychiatric disorder (adults)
* Any medical or social condition that in the opinion of the investigator will interfere with the study objectives or pose a risk to the study subject
* An employee (or first-degree relative of employee) of the Sponsor, the CRO, or any investigator or site personnel
* Female adult subjects who are pregnant or breast-feeding
* Adults with a recent history (within the past year) of alcohol or substance abuse.
* Toddlers who have already received a pentavalent booster (following the primary series).
* Toddlers with a family history of suspected primary immunodeficiency in first-degree relative.
* Toddlers who had a sibling die of likely sudden infant death syndrome (SIDS) or die suddenly and without apparent other cause or preceding illness in the first year of life.
* Toddlers with evidence of a clinically significant congenital abnormality as judged by the PI.
* Toddlers with evidence of fetal alcohol syndrome or maternal history of alcohol abuse during pregnancy

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Scott, MD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- KEMRI-Wellcome Trust Research Programme; Centre for Geographic Medicine Research - Coast, Kilifi, Kenya

RESULTS

PARTICIPANT FLOW:
Period: Received Vaccination 1
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo Low Dose | Adult Placebo High Dose | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo Low Dose | Toddler Placebo High Dose
Started | 12 | 12 | 12 | 12 | 50 | 50 | 50 | 50
Completed | 12 | 12 | 12 | 12 | 50 | 50 | 50 | 50
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Received Vaccination 2
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo Low Dose | Adult Placebo High Dose | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo Low Dose | Toddler Placebo High Dose
Started | 12 | 12 | 12 | 12 | 50 | 50 | 50 | 50
Completed | 11 | 11 | 12 | 12 | 50 | 49 | 50 | 49
Not Completed | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Had Immunology Data
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo Low Dose | Adult Placebo High Dose | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo Low Dose | Toddler Placebo High Dose
Started | 11 | 11 | 12 | 12 | 50 | 49 | 50 | 49
Completed | 11 | 11 | 12 | 12 | 50 | 49 | 49 (Subject received both vaccinations and attended last visit, but withdrew consent afterwards.) | 49
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo Low Dose | Adult Placebo High Dose | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo Low Dose | Toddler Placebo High Dose | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 50 | 50 | 50 | 50 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (7.04) | 30.8 (5.51) | 29.5 (6.74) | 27.6 (6.78) | 1.4 (0.25) | 1.4 (0.19) | 1.3 (0.21) | 1.4 (0.21) | 6.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 4 | 23 | 29 | 31 | 24 | 125
  Male | 8 | 7 | 7 | 8 | 27 | 21 | 19 | 26 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 12 | 12 | 12 | 50 | 50 | 50 | 50 | 248
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnic Group [Count of Participants; unit: Participants]
  Chonyi | 11 | 8 | 6 | 7 | 38 | 45 | 40 | 42 | 197
  Giriama | 1 | 2 | 4 | 2 | 9 | 5 | 9 | 5 | 37
  Luo | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 2 | 2 | 3 | 2 | 0 | 1 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Highest Grade of Reactogenicity Events in the Adult Cohort: Vaccination 1
Description: Solicited adverse events (AEs) were referred to as reactogenicity events (REs). Local REs included pain, induration/swelling, and erythema/redness at the injection site for adults; and pain/tenderness, redness, and induration/swelling for toddlers. Solicited systemic REs included cutaneous rash, headache, axillary fever/temperature, fatigue/malaise, and arthralgia/myalgia. Solicited REs were assessed for all subjects during the 60 minutes post-vaccination, daily for the first week, and at the clinic visit 1 week post-vaccination. Within the first week post-vaccination, fieldworkers visited the subject at home daily to assess and record solicited reactogenicity and determine whether the subject needed to be seen by the principal investigator (PI) for any medical condition or issue. Generally, grade 1 was no interference with activity, grade 2 was some interference with activity, and grade 3 was prevents daily activity. Grade 0 is equivalent to no event.
Time Frame: 7 days after the first dose (Day 7)
Measure: Count of Participants; unit: Participants
Groups:
- Adult Placebo: Two injections of normal saline with a 28 day interval between injections
  Placebo: Normal Saline
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo
Number analyzed (Participants) | 12 | 12 | 24
Participants
  Cutaneous Rash: Grade 0 | 11 | 12 | 22
  Cutaneous Rash: Grade 1 | 1 | 0 | 1
  Cutaneous Rash: Grade 2 | 0 | 0 | 1
  Cutaneous Rash: Grade 3 | 0 | 0 | 0
  Headache: Grade 0 | 11 | 8 | 19
  Headache: Grade 1 | 1 | 3 | 5
  Headache: Grade 2 | 0 | 1 | 0
  Headache: Grade 3 | 0 | 0 | 0
  Fatigue/Malaise: Grade 0 | 9 | 8 | 21
  Fatigue/Malaise: Grade 1 | 2 | 3 | 2
  Fatigue/Malaise: Grade 2 | 1 | 1 | 1
  Fatigue/Malaise: Grade 3 | 0 | 0 | 0
  Myalgia: Grade 0 | 10 | 8 | 23
  Myalgia: Grade 1 | 1 | 4 | 0
  Myalgia: Grade 2 | 1 | 0 | 1
  Myalgia: Grade 3 | 0 | 0 | 0
  Arthralgia: Grade 0 | 10 | 9 | 23
  Arthralgia: Grade 1 | 1 | 2 | 0
  Arthralgia: Grade 2 | 1 | 1 | 1
  Arthralgia: Grade 3 | 0 | 0 | 0
  Pain at Injection Site: Grade 0 | 2 | 0 | 17
  Pain at Injection Site: Grade 1 | 9 | 9 | 7
  Pain at Injection Site: Grade 2 | 1 | 2 | 0
  Pain at Injection Site: Grade 3 | 0 | 1 | 0
  Swelling/Hardness at injection site: Grade 0 | 12 | 10 | 24
  Swelling/Hardness at injection site: Grade 1 | 0 | 0 | 0
  Swelling/Hardness at injection site: Grade 2 | 0 | 2 | 0
  Swelling/Hardness at injection site: Grade 3 | 0 | 0 | 0

2. Primary Outcome: Highest Grade of Reactogenicity Events in the Adult Cohort: Vaccination 2
Description: Solicited adverse events (AEs) were referred to as reactogenicity events (REs). Local REs included pain, induration/swelling, and erythema/redness at the injection site for adults; and pain/tenderness, redness, and induration/swelling for toddlers. Solicited systemic REs included cutaneous rash, headache, axillary fever/temperature, fatigue/malaise, and arthralgia/myalgia. Solicited REs were assessed for all subjects during the 60 minutes post-vaccination, daily for the first week, and at the clinic visit 1 week post-vaccination. Within the first week post-vaccination, fieldworkers visited the subject at home daily to assess and record solicited reactogenicity and determine whether the subject needed to be seen by the principal investigator (PI) for any medical condition or issue. Generally, grade 1 was no interference with activity, grade 2 was some interference with activity, and grade 3 was prevents daily activity.
Time Frame: 7 days after the second dose (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo
Number analyzed (Participants) | 11 | 11 | 24
Participants
  Cutaneous Rash: Grade 0 | 11 | 11 | 22
  Cutaneous Rash: Grade 1 | 0 | 0 | 2
  Cutaneous Rash: Grade 2 | 0 | 0 | 0
  Cutaneous Rash: Grade 3 | 0 | 0 | 0
  Headache: Grade 0 | 10 | 10 | 19
  Headache: Grade 1 | 1 | 1 | 5
  Headache: Grade 2 | 0 | 0 | 0
  Headache: Grade 3 | 0 | 0 | 0
  Fatigue/Malaise: Grade 0 | 9 | 9 | 22
  Fatigue/Malaise: Grade 1 | 1 | 0 | 0
  Fatigue/Malaise: Grade 2 | 1 | 2 | 1
  Fatigue/Malaise: Grade 3 | 0 | 0 | 1
  Myalgia: Grade 0 | 10 | 10 | 24
  Myalgia: Grade 1 | 1 | 1 | 0
  Myalgia: Grade 2 | 0 | 0 | 0
  Myalgia: Grade 3 | 0 | 0 | 0
  Arthralgia: Grade 0 | 7 | 9 | 22
  Arthralgia: Grade 1 | 4 | 1 | 1
  Arthralgia: Grade 2 | 0 | 1 | 0
  Arthralgia: Grade 3 | 0 | 0 | 1
  Pain at Injection Site: Grade 0 | 4 | 2 | 15
  Pain at Injection Site: Grade 1 | 7 | 8 | 8
  Pain at Injection Site: Grade 2 | 0 | 1 | 1
  Pain at Injection Site: Grade 3 | 0 | 0 | 0
  Swelling/Hardness at injection site: Grade 0 | 11 | 10 | 24
  Swelling/Hardness at injection site: Grade 1 | 0 | 0 | 0
  Swelling/Hardness at injection site: Grade 2 | 0 | 1 | 0
  Swelling/Hardness at injection site: Grade 3 | 0 | 0 | 0
  Temperature: Grade 0 | 10 | 10 | 24
  Temperature: Grade 1 | 1 | 1 | 0
  Temperature: Grade 2 | 0 | 0 | 0
  Temperature: Grade 3 | 0 | 0 | 0

3. Primary Outcome: Highest Grade of Reactogenicity Events in the Toddler Cohort: Vaccination 1
Description: Solicited adverse events (AEs) were referred to as reactogenicity events (REs). Local REs included pain, induration/swelling, and erythema/redness at the injection site for adults; and pain/tenderness, redness, and induration/swelling for toddlers. Solicited systemic REs included cutaneous rash, axillary fever/temperature, drowsiness, irritability, and decreased appetite. Solicited REs were assessed for all subjects during the 60 minutes post-vaccination, daily for the first week, and at the clinic visit 1 week post-vaccination. Within the first week post-vaccination, fieldworkers visited the subject at home daily to assess and record solicited reactogenicity and determine whether the subject needed to be seen by the PI for any medical condition or issue. Generally, grade 1 was no interference with activity, grade 2 was some interference with activity, and grade 3 was prevents daily activity. Grade 0 is equivalent to no event.
Time Frame: 7 days after the first dose (Day 7)
Measure: Count of Participants; unit: Participants
Groups:
- Toddler Placebo: Two injections of normal saline with a 28 day interval between injections
  Placebo: Normal Saline
Arm/Group | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
Number analyzed (Participants) | 50 | 50 | 100
Participants
  Temperature: Grade 0 | 43 | 47 | 93
  Temperature: Grade 1 | 5 | 2 | 6
  Temperature: Grade 2 | 2 | 1 | 0
  Temperature: Grade 3 | 0 | 0 | 1
  Cutaneous Rash: Grade 0 | 46 | 44 | 91
  Cutaneous Rash: Grade 1 | 0 | 4 | 7
  Cutaneous Rash: Grade 2 | 4 | 2 | 2
  Cutaneous Rash: Grade 3 | 0 | 0 | 0
  Irritability: Grade 0 | 42 | 45 | 97
  Irritability: Grade 1 | 7 | 5 | 3
  Irritability: Grade 2 | 1 | 0 | 0
  Irritability: Grade 3 | 0 | 0 | 0
  Drowsiness: Grade 0 | 50 | 49 | 98
  Drowsiness: Grade 1 | 0 | 1 | 2
  Drowsiness: Grade 2 | 0 | 0 | 0
  Drowsiness: Grade 3 | 0 | 0 | 0
  Loss of appetite: Grade 0 | 41 | 48 | 95
  Loss of appetite: Grade 1 | 9 | 2 | 5
  Loss of appetite: Grade 2 | 0 | 0 | 0
  Loss of appetite: Grade 3 | 0 | 0 | 0
  Tenderness at injection site: Grade 0 | 29 | 41 | 94
  Tenderness at injection site: Grade 1 | 18 | 8 | 6
  Tenderness at injection site: Grade 2 | 3 | 1 | 0
  Tenderness at injection site: Grade 3 | 0 | 0 | 0
  Redness at injection site: Grade 0 | 48 | 46 | 94
  Redness at injection site: Grade 1 | 2 | 4 | 6
  Redness at injection site: Grade 2 | 0 | 0 | 0
  Redness at injection site: Grade 3 | 0 | 0 | 0
  Swelling/hardness at injection site: Grade 0 | 46 | 45 | 99
  Swelling/hardness at injection site: Grade 1 | 4 | 5 | 1
  Swelling/hardness at injection site: Grade 2 | 0 | 0 | 0
  Swelling/hardness at injection site: Grade 3 | 0 | 0 | 0

4. Primary Outcome: Highest Grade of Reactogenicity Events in the Toddler Cohort: Vaccination 2
Description: as for outcome 3
Time Frame: 7 days after the second dose (Day 35)
Measure: Count of Participants; unit: Participants
Arm/Group | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
Number analyzed (Participants) | 50 | 50 | 100
Participants
  Temperature: Grade 0 | 42 | 41 | 80
  Temperature: Grade 1 | 5 | 6 | 11
  Temperature: Grade 2 | 3 | 2 | 8
  Temperature: Grade 3 | 0 | 1 | 1
  Cutaneous Rash: Grade 0 | 45 | 46 | 93
  Cutaneous Rash: Grade 1 | 4 | 4 | 6
  Cutaneous Rash: Grade 2 | 1 | 0 | 1
  Cutaneous Rash: Grade 3 | 0 | 0 | 0
  Irritability: Grade 0 | 30 | 32 | 61
  Irritability: Grade 1 | 18 | 17 | 36
  Irritability: Grade 2 | 2 | 1 | 3
  Irritability: Grade 3 | 0 | 0 | 0
  Drowsiness: Grade 0 | 48 | 49 | 89
  Drowsiness: Grade 1 | 2 | 1 | 9
  Drowsiness: Grade 2 | 0 | 0 | 2
  Drowsiness: Grade 3 | 0 | 0 | 0
  Loss of appetite: Grade 0 | 36 | 36 | 78
  Loss of appetite: Grade 1 | 10 | 14 | 20
  Loss of appetite: Grade 2 | 4 | 0 | 2
  Loss of appetite: Grade 3 | 0 | 0 | 0
  Tenderness at injection site: Grade 0 | 30 | 36 | 75
  Tenderness at injection site: Grade 1 | 13 | 12 | 21
  Tenderness at injection site: Grade 2 | 6 | 2 | 2
  Tenderness at injection site: Grade 3 | 1 | 0 | 2
  Redness at injection site: Grade 0 | 46 | 49 | 97
  Redness at injection site: Grade 1 | 4 | 1 | 3
  Redness at injection site: Grade 2 | 0 | 0 | 0
  Redness at injection site: Grade 3 | 0 | 0 | 0
  Swelling/hardness at injection site: Grade 0 | 47 | 46 | 93
  Swelling/hardness at injection site: Grade 1 | 0 | 4 | 4
  Swelling/hardness at injection site: Grade 2 | 3 | 0 | 3
  Swelling/hardness at injection site: Grade 3 | 0 | 0 | 0

5. Secondary Outcome: Immunoglobulin G (IgG) Antibody Geometric Mean Concentration Against Pneumococcal Proteins
Description: Proteins were measured on the Meso Scale Discovery (MSD) platform using an an electrochemiluminescence detection assay. Units were arbitrary.
Time Frame: Baseline and 12 weeks after vaccination 2 (Day 0 and Day 112)
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo Low Dose | Adult Placebo High Dose | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo Low Dose | Toddler Placebo High Dose
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 50 | 49 | 49 | 49
arbitrary units
  L460D: Baseline | 642.5 [370.6 to 1113.8] | 804.6 [462.2 to 1400.7] | 614.4 [484.5 to 779.2] | 1022.3 [755.4 to 1383.5] | 267.7 [199.2 to 359.6] | 326.8 [258.5 to 413.1] | 197.4 [158.2 to 246.4] | 330.6 [253.9 to 430.5]
  L460D: Post-vaccination 2 | 1004.1 [608.8 to 1656.1] | 1294.2 [781.3 to 2143.7] | 620.3 [455.0 to 845.6] | 943.0 [658.4 to 1350.6] | 422.1 [313.0 to 569.1] | 563.6 [442.0 to 718.7] | 262.3 [206.6 to 332.9] | 389.6 [294.7 to 515.2]
  PspA-Fam1: Baseline | 1555.7 [791.5 to 3057.8] | 1342.1 [689.9 to 2610.7] | 2145.3 [1476.3 to 3117.4] | 2837.2 [1792.5 to 4490.7] | 197 [123.2 to 315.1] | 358 [264.0 to 485.4] | 230.3 [164.4 to 322.6] | 414.4 [278.1 to 617.4]
  PspA-Fam1: Post-vaccination 2 | 3344.5 [1868.9 to 5985.2] | 2684.4 [1475.7 to 4883.1] | 2071.8 [1345.9 to 3189.3] | 2588.5 [1558.8 to 4298.5] | 326.2 [211.7 to 502.6] | 593.8 [433.9 to 812.6] | 315.1 [231.5 to 429.0] | 560.4 [376.9 to 833.3]
  PhtD: Baseline | 736.6 [441.9 to 1227.6] | 942.3 [506.3 to 1754.0] | 655.7 [453.0 to 949.1] | 619.5 [456.2 to 841.4] | 671.3 [498.1 to 904.6] | 713.2 [537.6 to 946.3] | 644.1 [473.1 to 876.7] | 775.8 [563.6 to 1068.0]
  PhtD: Post-vaccination 2 | 842.5 [497.8 to 1426.0] | 923.3 [530.6 to 1606.6] | 663.8 [451.4 to 976.2] | 592 [422.0 to 830.6] | 870.3 [655.2 to 1156.1] | 1064.5 [826.7 to 1370.9] | 776.3 [595.7 to 1011.8] | 922.7 [695.7 to 1223.6]
  BCH0785: Baseline | 593.8 [349.4 to 1008.9] | 562.3 [299.5 to 1055.7] | 1214.5 [729.7 to 2021.3] | 790.1 [425.3 to 1467.5] | 287.4 [208.0 to 397.1] | 389.3 [288.8 to 524.9] | 237.1 [168.9 to 332.7] | 346.6 [246.7 to 487.1]
  BCH0785: Post-vaccination 2 | 713.5 [410.0 to 1241.6] | 640.6 [383.3 to 1070.8] | 1205 [730.8 to 1986.9] | 747.9 [421.2 to 1328.2] | 398 [284.8 to 556.1] | 627.8 [467.7 to 842.7] | 301.8 [219.1 to 415.8] | 367.4 [261.9 to 515.2]
  StkP: Baseline | 524.6 [255.5 to 1076.8] | 917.6 [484.9 to 1736.2] | 1270.6 [819.5 to 1970.0] | 973.3 [539.9 to 1754.7] | 192 [136.8 to 269.5] | 218.9 [160.4 to 298.8] | 153.6 [113.1 to 208.6] | 197 [141.8 to 273.8]
  StkP: Post-vaccination 2 | 701.1 [343.2 to 1432.3] | 1209.4 [729.7 to 2004.3] | 1329.5 [859.3 to 2056.9] | 907.7 [512.9 to 1606.2] | 346 [245.4 to 487.8] | 409 [309.3 to 540.9] | 199.1 [147.2 to 269.3] | 211.6 [152.0 to 294.6]
  PcpA: Baseline | 1099.7 [629.2 to 1922.2] | 967 [536.3 to 1743.6] | 1240.7 [874.6 to 1760.1] | 1053.8 [784.5 to 1415.6] | 505.8 [324.9 to 787.4] | 431.9 [286.1 to 652.0] | 635.4 [398.9 to 1011.9] | 506.1 [322.7 to 793.8]
  PcpA: Post-vaccination 2 | 1094.6 [608.8 to 1968.0] | 820.8 [499.0 to 1350.0] | 1259.7 [870.2 to 1823.6] | 972.3 [741.6 to 1274.9] | 611.3 [395.0 to 946.0] | 580.6 [378.2 to 891.5] | 778.3 [489.2 to 1238.4] | 737.5 [493.1 to 1102.8]
  SPWCV: Baseline | 938.2 [787.3 to 1118.1] | 886.3 [618.9 to 1269.3] | 893.5 [792.2 to 1007.7] | 742 [587.7 to 936.8] | 495.2 [433.5 to 565.8] | 544.9 [463.3 to 640.8] | 488.3 [429.7 to 554.9] | 590.8 [516.6 to 675.7]
  SPWCV: Post-vaccination 2 | 1042.2 [853.0 to 1273.3] | 954.9 [714.7 to 1275.9] | 930.6 [785.9 to 1101.9] | 698.9 [562.7 to 868.1] | 636.8 [555.1 to 730.5] | 688.8 [605.0 to 784.3] | 562.1 [499.8 to 632.2] | 654.5 [570.9 to 750.4]
  PiuA: Baseline | 659.7 [372.6 to 1167.9] | 796.1 [509.9 to 1243.0] | 1554.8 [848.3 to 2849.5] | 1223.9 [625.0 to 2396.6] | 811.6 [638.3 to 1032.0] | 917.7 [735.1 to 1145.7] | 665.4 [507.6 to 872.2] | 888 [677.2 to 1164.5]
  PiuA: Post-vaccination 2 | 1001.9 [496.4 to 2022.1] | 1049.7 [655.9 to 1680.0] | 1540.4 [843.2 to 2813.9] | 1214.3 [621.0 to 2374.4] | 1091.9 [857.6 to 1390.3] | 1343.2 [1044.9 to 1726.6] | 809 [639.0 to 1024.4] | 899 [681.2 to 1186.4]
  PiaA: Baseline | 1313.4 [674.9 to 2556.0] | 1462.5 [788.2 to 2713.8] | 1620.3 [1061.7 to 2472.9] | 1611.4 [1027.4 to 2527.5] | 560.6 [404.0 to 778.0] | 662.8 [527.2 to 833.1] | 571.4 [431.4 to 756.8] | 626.5 [473.7 to 828.4]
  PiaA: Post-vaccination 2 | 1768.8 [850.6 to 3678.1] | 1802.5 [1036.0 to 3136.3] | 1540 [958.0 to 2475.5] | 1638.8 [1018.4 to 2636.9] | 743.6 [537.3 to 1029.1] | 904.3 [703.5 to 1162.2] | 647.6 [505.0 to 830.4] | 640.5 [484.1 to 847.4]

6. Secondary Outcome: Immunoglobulin G (IgG) Antibody Geometric Mean Fold Change Against Pneumococcal Proteins
Description: Between baseline and 28 days after vaccination 2. Proteins were measured on the Meso Scale Discovery (MSD) platform using an an electrochemiluminescence detection assay.
Time Frame: Baseline and 12 weeks after vaccination 2 (Day 0 and Day 112)
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
Number analyzed (Participants) | 11 | 11 | 24 | 50 | 49 | 98
fold change
  L460D | 1.56 [1.28 to 1.91] | 1.61 [1.24 to 2.09] | 0.97 [0.88 to 1.05] | 1.58 [1.35 to 1.84] | 1.72 [1.45 to 2.05] | 1.25 [1.11 to 1.41]
  PspA-Fam1 | 2.15 [1.47 to 3.14] | 2.00 [1.18 to 3.38] | 0.94 [0.87 to 1.02] | 1.66 [1.34 to 2.04] | 1.66 [1.36 to 2.03] | 1.36 [1.11 to 1.67]
  PhtD | 1.14 [0.96 to 1.36] | 0.98 [0.82 to 1.16] | 0.98 [0.91 to 1.06] | 1.30 [1.11 to 1.51] | 1.49 [1.31 to 1.70] | 1.20 [1.07 to 1.34]
  BCH0785 | 1.20 [1.02 to 1.42] | 1.14 [0.77 to 1.68] | 0.97 [0.90 to 1.04] | 1.38 [1.15 to 2.15] | 1.87 [1.53 to 2.28] | 1.18 [1.06 to 1.32]
  StkP | 1.34 [1.10 to 1.62] | 1.32 [0.98 to 1.77] | 0.99 [0.92 to 1.06] | 1.80 [1.51 to 2.15] | 1.87 [1.53 to 2.28] | 1.18 [1.06 to 1.32]
  PcpA | 1.00 [0.87 to 1.14] | 0.85 [0.65 to 1.11] | 0.97 [0.90 to 1.05] | 1.21 [0.98 to 1.49] | 1.34 [1.06 to 1.70] | 1.34 [1.11 to 1.61]
  SPWCV | 1.11 [0.93 to 1.33] | 1.08 [0.88 to 1.32] | 0.99 [0.91 to 1.07] | 1.29 [1.13 to 1.47] | 1.26 [1.12 to 1.43] | 1.12 [1.05 to 1.20]
  PiuA | 1.52 [1.17 to 1.97] | 1.32 [0.84 to 2.08] | 0.99 [0.93 to 1.06] | 1.35 [1.12 to 1.62] | 1.46 [1.22 to 1.76] | 1.11 [0.98 to 1.25]
  PiaA | 1.35 [1.10 to 1.65] | 1.23 [0.99 to 1.54] | 0.98 [0.90 to 1.08] | 1.33 [1.14 to 1.55] | 1.36 [1.15 to 1.62] | 1.08 [0.94 to 1.24]

7. Secondary Outcome: Number of Subjects With Immunoglobulin G (IgG) Seroresponse
Description: as for outcome 6
Time Frame: Baseline and 12 weeks after vaccination 2 (Day 0 and Day 112)
Measure: Count of Participants; unit: Participants
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
Number analyzed (Participants) | 11 | 11 | 24 | 50 | 49 | 98
Participants
  L460D: <2 fold rise | 9 | 9 | 24 | 34 | 33 | 78
  L460D: Between 2 and 3 fold rise | 2 | 0 | 0 | 12 | 11 | 13
  L460D: Between 3 and 4 fold rise | 0 | 2 | 0 | 2 | 1 | 6
  L460D: ≥4 fold rise | 0 | 0 | 0 | 2 | 4 | 1
  PspA-Fam1: <2 fold rise | 6 | 9 | 24 | 31 | 30 | 72
  PspA-Fam1: Between 2 and 3 fold rise | 2 | 0 | 0 | 11 | 12 | 6
  PspA-Fam1: Between 3 and 4 fold rise | 0 | 0 | 0 | 5 | 3 | 2
  PspA-Fam1: ≥4 fold rise | 3 | 2 | 0 | 3 | 4 | 18
  PhtD: <2 fold rise | 11 | 11 | 24 | 37 | 39 | 78
  PhtD: Between 2 and 3 fold rise | 0 | 0 | 0 | 11 | 4 | 17
  PhtD: Between 3 and 4 fold rise | 0 | 0 | 0 | 2 | 6 | 2
  PhtD: ≥4 fold rise | 0 | 0 | 0 | 0 | 0 | 1
  BCH0785: <2 fold rise | 11 | 10 | 24 | 36 | 33 | 81
  BCH0785: Between 2 and 3 fold rise | 0 | 1 | 0 | 7 | 6 | 6
  BCH0785: Between 3 and 4 fold rise | 0 | 0 | 0 | 4 | 4 | 5
  BCH0785: ≥4 fold rise | 0 | 0 | 0 | 3 | 6 | 6
  StkP: <2 fold rise | 9 | 10 | 24 | 25 | 27 | 78
  StkP: Between 2 and 3 fold rise | 2 | 0 | 0 | 16 | 12 | 15
  StkP: Between 3 and 4 fold rise | 0 | 0 | 0 | 1 | 5 | 3
  StkP: ≥4 fold rise | 0 | 1 | 0 | 8 | 5 | 2
  PcpA: <2 fold rise | 11 | 11 | 24 | 44 | 33 | 69
  PcpA: Between 2 and 3 fold rise | 0 | 0 | 0 | 1 | 7 | 13
  PcpA: Between 3 and 4 fold rise | 0 | 0 | 0 | 3 | 5 | 7
  PcpA: ≥4 fold rise | 0 | 0 | 0 | 2 | 4 | 9
  SPWCV: <2 fold rise | 11 | 11 | 24 | 43 | 45 | 95
  SPWCV: Between 2 and 3 fold rise | 0 | 0 | 0 | 6 | 2 | 3
  SPWCV: Between 3 and 4 fold rise | 0 | 0 | 0 | 0 | 1 | 0
  SPWCV: ≥4 fold rise | 0 | 0 | 0 | 1 | 1 | 0
  PiuA: <2 fold rise | 9 | 9 | 24 | 40 | 37 | 82
  PiuA: Between 2 and 3 fold rise | 1 | 2 | 0 | 6 | 6 | 11
  PiuA: Between 3 and 4 fold rise | 1 | 0 | 0 | 0 | 3 | 4
  PiuA: ≥4 fold rise | 0 | 0 | 0 | 4 | 3 | 1
  PiaA: <2 fold rise | 9 | 10 | 24 | 43 | 38 | 89
  PiaA: Between 2 and 3 fold rise | 2 | 1 | 0 | 3 | 5 | 3
  PiaA: Between 3 and 4 fold rise | 0 | 0 | 0 | 1 | 4 | 4
  PiaA: ≥4 fold rise | 0 | 0 | 0 | 3 | 2 | 2

8. Primary Outcome: Number of Adverse Events (AE), by Relation to Vaccine and Seriousness
Description: Only treatment-emergent adverse events (TEAEs) were included in the analysis; adverse events (AEs) that were not TEAEs were to have been listed.
Time Frame: 112 days
Measure: Number; unit: adverse events
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
Number analyzed (Participants) | 12 | 12 | 24 | 50 | 50 | 100
adverse events
  Serious : Related | 0 | 0 | 0 | 0 | 0 | 2
  Serious : Not related | 0 | 0 | 0 | 3 | 2 | 3
  Non-serious : Related | 0 | 0 | 0 | 0 | 2 | 1
  Non-serious : Not related | 18 | 21 | 39 | 148 | 80 | 253

ADVERSE EVENTS:
Time Frame: 112 days from receipt of first vaccination
Arm/Group | Adult 0.6mg PATH-wSP | Adult 1.0 mg PATH-wSP | Adult Placebo | Toddler 0.6mg PATH-wSP | Toddler 1.0 mg PATH-wSP | Toddler Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 0/50 | 0/50 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 2/50 | 1/50 | 5/100
Other Adverse Events (participants affected / at risk) | 9/12 | 9/12 | 20/24 | 45/50 | 44/50 | 87/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult 0.6mg PATH-wSP (N=12) | Adult 1.0 mg PATH-wSP (N=12) | Adult Placebo (N=24) | Toddler 0.6mg PATH-wSP (N=50) | Toddler 1.0 mg PATH-wSP (N=50) | Toddler Placebo (N=100)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Pneumococcal bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult 0.6mg PATH-wSP (N=12) | Adult 1.0 mg PATH-wSP (N=12) | Adult Placebo (N=24) | Toddler 0.6mg PATH-wSP (N=50) | Toddler 1.0 mg PATH-wSP (N=50) | Toddler Placebo (N=100)
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 9 | 27 | 3 | 23
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 11 | 2 | 11
Tonsillitis (Infections and infestations) | 1 | 1 | 2 | 3 | 4 | 7
Conjunctivitis (Infections and infestations) | 0 | 1 | 2 | 3 | 6 | 8
Malaria (Infections and infestations) | 1 | 0 | 2 | 3 | 1 | 6
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 20 | 23 | 47
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 1 | 0 | 0 | 3 | 3 | 11
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Helminthic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 4
Mastitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 13 | 7 | 11
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 5
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess of eyelid (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Septic rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0
Toothache (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 13 | 6 | 20
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 2 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 4
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2
Greenstick fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 7 | 13
Vaccination site induration (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02543892/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02543892/SAP_001.pdf